CLINICAL TRIAL: NCT01603251
Title: A Double Blind Randomized Controlled Trial of Artemether-Lumefantrine Alone and in Combination With Ivermectin to Reduce Post-Treatment Malaria Transmission
Brief Title: Trial of Artemether-Lumefantrine Alone and in Combination With Ivermectin to Reduce Post-Treatment Malaria Transmission
Acronym: ACTIVE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Radboud University Medical Center (Other); Centre national de recherche et de formation sur le paludisme (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACTIVE
Record Dates: First submitted 2012-05-16; First posted 2012-05-22 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Malaria
Keywords: transmission; anopheles
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination; Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Artemether-Lumefantrine (Active Comparator)
  Interventions: Drug: Artemether-lumefantrine combination
- Artemether-Lumefantrine + single dose Ivermectin (Experimental)
  Interventions: Drug: Artemether-lumefantrine combination + single dose Ivermectin
- Artemether-Lumefantrine + repeated dose Ivermectin (Experimental)
  Interventions: Drug: Artemether-lumefantrine combination + repeated dose Ivermectin

INTERVENTIONS:
Drug: Artemether-lumefantrine combination — Artemether-Lumefantrine (AL)combination; a placebo is given together with the first and fifth dose of AL
  Arms: Artemether-Lumefantrine
Drug: Artemether-lumefantrine combination + single dose Ivermectin — Artemether-lumefantrine (AL) combination + Ivermectin (200ug/kg) given once together with the first dose of AL. A placebo is given together with the fifth dose of AL.
  Arms: Artemether-Lumefantrine + single dose Ivermectin
Drug: Artemether-lumefantrine combination + repeated dose Ivermectin — Artemether-lumefantrine (AL) combination + Ivermectin (200ug/kg) given together with the first and fifth dose of AL.
  Arms: Artemether-Lumefantrine + repeated dose Ivermectin

SUMMARY:
The purpose of this study is to determine the safety and impact of ivermectin, administered as single or repeated dose, in combination with artemether-lumefantrine in reducing the proportion of mosquitoes that survive and become infected after feeding on a blood meal from a malaria-infected individual.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatically infected individuals with any P. falciparum parasite density

Exclusion Criteria:

* age < 15 years or > 25 years
* malaria parasite density ≥ 10,000 parasites/µL
* clinical symptoms indicating severe malaria
* axillary temperature ≥ 37.5°C
* Body Mass Index (BMI) below 18 or above 32 kg/m2
* haemoglobin concentration below 11 g/dL
* taken ivermectin in the last three months
* Loa loa as assessed by questionnaire, clinical examination and parasitological assessments
* for women: pregnancy or lactation
* known hypersensitivity to AL or IVM
* history and/or symptoms indicating chronic illness
* current use of tuberculosis or anti-retroviral medication
* unable to give written informed consent
* unwillingness to participate in two membrane feeding assays
* travel history to Angola, Cameroon, Chad, Central African Republic, Congo, DR Congo, Equatorial Guinea, Ethiopia, Gabon, Nigeria and Sudan. If a potential participant has ever visited one or more of these countries, he or she will not be eligible for enrolment.
* history of cardiovascular disease.
* taking drugs that are known to influence cardiac function and to prolong QTc interval, such as class IA and III: neuroleptics, antidepressant agents, certain antibiotics including some agents of the following classes - macrolides, fluoroquinolones, imidazole, and triazole antifungal agents, certain non-sedating antihistaminics (terfenadine, astemizole) and cisapride.
* known disturbances of electrolyte balance, e.g. hypokalaemia or hypomagnesaemia.
* taking drugs which may be metabolized by cytochrome enzyme CYP2D6 (e.g., flecainide, metoprolol, imipramine, amitriptyline, clomipramine).

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety | 8 days
  The number of adverse events; number of participants with abnormal haemoglobin, biochemistry or full blood count values

SECONDARY OUTCOMES:
Mosquitocidal activity | feeding experiments performed up to 8 days after enrolment; survival of mosquitoes determined up to day 10 after feeding
  Daily mortality rates of (malaria-infected) Anopheles gambiae s.s. and An. funestus mosquitoes after taking a blood meal 1, 3 or 7 days after initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Teun Bousema, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Centre National de Recherche et de Formation sur le Paludisme, Ouagadougou, Burkina Faso